CLINICAL TRIAL: NCT04535206
Title: The Relationship Between the Lack of Plasma Antithrombin Ⅲ, Protein C, Protein S Activity and Peripherally Inserted Central Catheter Related Thrombosis
Brief Title: The Relationship Between the Lack of AT-Ⅲ, PC, PS Activity and PICC-related Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-005
Record Dates: First submitted 2020-08-23; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Central Venous Catheter Thrombosis
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With AT-Ⅲ, PC, PS activity decreased: Any decreased in AT-Ⅲ, PC, PS activity before catheter intubation is regarded as the exposure group
  Interventions: Diagnostic Test: Venous blood collecting and test and ultrasound screening
- AT-Ⅲ, PC, PS activity are at normal value: The activities of AT-Ⅲ, PC and PS are all at normal values before catheter intubation
  Interventions: Diagnostic Test: Venous blood collecting and test and ultrasound screening

INTERVENTIONS:
Diagnostic Test: Venous blood collecting and test and ultrasound screening — To collect the venous blood samples before the PICC catheterization, and perform ultrasound examination before and after the catheterization at the specified time point in follow-up.

SUMMARY:
PICC related venous thrombosis (PICC-RVT) is one of the common complications of PICC and the main cause of unplanned extubation. Effectively identifying the risk of PICC-RVT in patients and preventing PICC-RVT are of great clinical significance. There are many studies on the risk factors of VTE at home and abroad, and there are also many studies on the risk assessment of PICC catheter-related thrombosis, mostly focusing on sociodemographic data, comorbidities, and intubation related factors, while the research on laboratory related indicators is limited It involves D-dimer, white blood cell count (WBC), platelet count (PLT), etc., but its specificity or positive predictive value is not high, and there is no reliable biomarker report. Studies have shown that the decrease or lack of AT-Ⅲ, PC, PS activity is one of the mechanisms of hypercoagulable state in patients with cancer, and may be a biomarker of thrombosis. Many retrospective studies have also shown that the activities of AT-Ⅲ, PC, and PS are related to the occurrence and recurrence of VTE and DVT. The pathogenesis is mainly anticoagulant protein defect or decreased expression. However, when PICC is implanted in patients with AT-Ⅲ, PC and PS activity defects, whether PICC indwelling will become a predisposing factor of thrombosis is not yet known. Therefore, the purpose of this study is to understand the rate of anticoagulant protein deficiency in patients with tumor PICC-RVT, and to prospectively explore the correlation between the lack of AT-Ⅲ, PC, and PS activities and PICC-RVT, and to provide targeted preventive interventions for PICC-RVT patients Scientific basis.

DETAILED DESCRIPTION:
A prospective study showed that a mild reduction in AT levels (70%-80%) was associated with the recurrence of no incentive VTE. Subsequent studies defined mild AT deficiency as less than the 5th percentile of the normal range to further verify that mild AT deficiency is a risk factor for VTE recurrence. Many retrospective studies have also shown that the activities of AT-Ⅲ, PC and PS are related to the occurrence and recurrence of VTE and DVT. Taking the lower limit of the normal reference value as the criterion for judging the lack of anticoagulant protein activity, Zhu Tienan et al. found that the lack of activity of AT, PC, and PS in normal people were 1.15%, 1.49%, and 2.29%, respectively. Fang Biqian et al. found 277 cases of VTE. Among the cases found that the lack of activity of AT, PC, and PS were 16.00%, 17.45%, and 17.09%, respectively. That is, the lack of activity of the three anticoagulant proteins in VTE patients was about 10 times higher than that of normal people. Chinese scholars from Taiwan, Hong Kong and Shanghai also found that the total lack of three anticoagulant proteins of AT-Ⅲ, PC and PS exceeds 15% in Western countries, suggesting that the etiological composition of venous thromboembolism in the Chinese population may be similar to that of Western countries. Different, reflecting that anticoagulant protein deficiency plays an important role in the pathogenesis of VTE patients in China. Compared with factor V Leiden mutation and prothrombin 20210A mutation, the most common thrombosis in Asian population is antithrombin Ⅲ (AT-Ⅲ), protein C (protein C, PC) and protein S (protein S, PS), etc. Defects of anticoagulant protein. When the hypercoagulable state caused by anticoagulant protein deficiency is induced by certain risk factors for thrombosis, such as pregnancy, oral contraceptives, fractures, long-term immobilization, etc., it can lead to the occurrence of VTE. When PICC is implanted in patients with AT-Ⅲ, PC and PS activity defects, whether PICC indwelling will become a predisposing factor of thrombosis is not yet known.

It has been reported that the severity of CVC-related thrombosis in patients with AT-Ⅲ deficiency after CVC catheterization is higher than that of the normal group. Nowak-Göttl et al. showed that PC and PS genetic defects are related to catheterization in children Thrombosis plays an important role. In 2016, a systematic review showed that the risk of DVT related to more than one anticoagulant defect increased by 3.20 times. PC defects can increase the incidence of CVC-related DVT in children. Our preliminary study of this subject found that the lack of anticoagulant protein in PICC-RVT patients was higher than that in non-PICC-RVT patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; Patients with solid tumors in line with the indications for catheterization; PICC Intubation and maintenance in this hospital; Expected catheter indwelling time ≥8 weeks; Willing to cooperate with this study and sign an informed consent

Exclusion Criteria:

* With Pregnant; with mental diseases who cannot cooperate; Incomplete clinical data; The catheter tip position is not in the best position or the catheter-to-venous ratio ≥45% (vascular diameter≤2.93 mm); Have thrombosis in 3 months before intubation; Be undergoing thrombolysis or anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumors and have PICC intubation in this tertiary hospital are recruited in order.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PICC-RVT | 8 weeks
  The incidence of PICC-related thrombosis

SECONDARY OUTCOMES:
The incidence of other VTE | Through study completion, an average of 1 year
  The incidence of other VTE not related to PICC

CONTACTS AND LOCATIONS:
Overall Officials: Jingfen Jin, Master, Study Director — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China